CLINICAL TRIAL: NCT02482701
Title: An International, Multicenter, Prospective, Post Market Registry Using a New Device for Endoscopic Resection of Early Neoplasia in Barrett's Esophagus
Brief Title: The Captivator EMR Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 91038126
Record Dates: First submitted 2015-06-15; First posted 2015-06-26 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Barrett's Esophagus
Keywords: EMR; EAC; Barrett's Neoplasia; Multiband Mucosectomy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Captivator™ EMR — The Captivator ™ EMR Device is indicated for endoscopic mucosal resection (EMR) in the upper gastrointestinal (GI) tract.

SUMMARY:
To confirm performance of the Captivator™ EMR device for resection of early neoplasia in Barrett's Esophagus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Barrett's esophagus with a visible abnormality confirmed upon prior endoscopy. A visible abnormality is described as meeting one or more of the following definitions:

   * Lesion is detected as visible based on white light imaging with any macroscopic appearance according to the Paris Classification and is also endoscopically resectable.
   * Lesion is detected by narrow band imaging (NBI), but without any other specific characteristics for a visible lesion.
   * Lesion is confirmed to contain high grade dysplasia and/or carcinoma upon prior biopsy.
3. Subject is scheduled for endoscopic resection of present neoplasia
4. Subject is amenable to EMR with no suspicion of submucosal invasion, based on the macroscopic appearance and/or endosonography upon earlier endoscopy.
5. Subject is taking PPI (Proton Pump Inhibitor) BID (Twice Daily) 40 mg (or equivalent dosage).
6. Subject is willing to participate, fully understands the content of the informed consent form, and signs the informed consent form.

Exclusion Criteria:

1. Subject has previously undergone endoscopic therapy for esophageal neoplasia, including (but not limited to) cryospray therapy, laser treatment, photodynamic therapy, endoscopic mucosal resection, radiofrequency ablation, argon plasma coagulation or radiotherapy.
2. Presence of esophageal stenosis preventing passage of a therapeutic gastroscope.
3. Endoscopically visible scarring by any cause of the intended treatment zone.
4. Esophageal varices.
5. Subject has known or suspected esophageal perforation.
6. Coagulation disorders or anti-coagulant therapy which cannot be discontinued (aspirin allowed).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Barrett's Esophagus patients with early neoplasia.
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Successful endoscopic resection defined as complete resection of the delineated area, including all delineation markings, in a single procedure. | Procedure
  Successful resection is assessed during the EMR procedure

SECONDARY OUTCOMES:
Number of resections per procedure | Procedure
  The number of resection per procedure is assessed during the EMR Procedure
Total procedure time | Procedure
  Total procedure time is assessed during the EMR procedure
Seriousness and severity of adverse events related to the Captivator™ EMR device or procedure | Procedure through 30 days post EMR procedure
  Study subjects will have follow-up visits after the EMR procedure during which the occurrence of adverse events related to the Captivator EMR procedure or device will be assessed. These visits will occur at the following time points:
  * Immediately following the EMR procedure (Post procedure evaluation)
  * 48 hour telephone call
  * 30 day telephone call
  * Unscheduled clinic visits will be performed in-between protocol required follow-up, as necessary.
  Once the 30 day phone call is complete, the subject will have completed the study.
Accessory devices used during the procedure for complication management | Procedure
  Accessory device use is assessed during the EMR procedure
Ability to endoscopically manage complications without the need for additional interventions | Procedure
  Endoscopic management of complications is assessed during the EMR procedure
Accessory devices used to complete the resection procedure | Procedure
  Accessory devices used to complete resection is assessed during the EMR procedure
Histopathology | Post Procedure
  Histopathology of resection specimens is performed per standard of practice at each participating study center. Results are expected within approximately 7 days of the EMR procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bergman, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (13):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
- University Hospital Leuven, Leuven, Belgium
- St. Michael's Hospital, Toronto, Ontario, Canada
- Germany (2):
  - Krankenhaus Barmherzige Bruder, Regensburg, Bavaria
  - EVK Krankenhaus, Düsseldorf
- Netherlands (4):
  - Academic Medical Center, Amsterdam, AZ
  - Catharina Hospital, Eindhoven, EJ
  - St. Antonius Hospital, Nieuwgein, NL
  - Erasmus MC - University Medical Center, Rotterdam
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - University College Hospital, London
  - Nottingham Digestive Disease Centre, NIHR, Nottingham

REFERENCES:
- [Derived] Pouw RE, Beyna T, Belghazi K, Koch AD, Schoon EJ, Haidry R, Weusten BL, Bisschops R, Shaheen NJ, Wallace MB, Marcon N, Heise-Ginsburg R, Gotink AW, Wang KK, Leggett CL, Ortiz-Fernandez-Sordo J, Ragunath K, DiPietro M, Pech O, Neuhaus H, Bergman JJ. A prospective multicenter study using a new multiband mucosectomy device for endoscopic resection of early neoplasia in Barrett's esophagus. Gastrointest Endosc. 2018 Oct;88(4):647-654. doi: 10.1016/j.gie.2018.06.030. Epub 2018 Jul 6. PMID 30220300